CLINICAL TRIAL: NCT00519129
Title: Magnetic Endoscopic Imaging Versus Standard Colonoscopy in a Routine Colonoscopy Setting: A Randomised Controlled Trial
Brief Title: Improving Quality of Colonoscopy Using a 3D-imager
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sorlandet Hospital HF, Sorlandet Hospital HF
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SSHF-Colon-1
Record Dates: First submitted 2007-08-21; First posted 2007-08-22 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-08

CONDITIONS: Pain During Colonoscopy
Keywords: Pain; Patient satisfaction
MeSH Terms: conditions — Pain; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: 3D-imager — 3D-imager vs fluoroscopy during coloscopy
  Other Names: Skopguide

SUMMARY:
Coloscopy may be a painful procedure for the patient. This is due to a loop-formation of the coloscope. A 3D-real time imager produced by Olympus creates a real-time image of the scope while a traditional fluoroscopy device will only show instant pictures. We want to investigate whether the 3D-imager causes the patient less pain and is more time consuming than ordinary fluoroscopy

DETAILED DESCRIPTION:
Results published in Holme et.al. Gastrointestinal Endoscopy 2011;73:1215-1222.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for coloscopy on an out-patient basis

Exclusion Criteria:

* Pregnancy
* Pacemaker
* Lack of ability to understand information given
* Prior resection of the colon/rectum
* Demanding analgetics prior to start of procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2007-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
pain during coloscopy | instant
Time used to reach the coecum | instant

SECONDARY OUTCOMES:
coecum-intubation rate | instant
level achieved when the coecum can not be reached | instant
Need for assistance by a colleague | instant
Need for analgetics | instant
Pain during the first 24 hours after coloscopy | 24 hours
Polyp detection rate | instant

CONTACTS AND LOCATIONS:
Overall Officials: Geir S Hoff, PhD, Study Director
Locations (1):
- Sorlandet Sykehus HF, Kristiansand, Norway

REFERENCES:
- [Derived] Holme O, Hoie O, Matre J, Stallemo A, Garborg K, Hasund A, Wiig H, Hoff G, Bretthauer M. Magnetic endoscopic imaging versus standard colonoscopy in a routine colonoscopy setting: a randomized, controlled trial. Gastrointest Endosc. 2011 Jun;73(6):1215-22. doi: 10.1016/j.gie.2011.01.054. Epub 2011 Apr 8. PMID 21481862